CLINICAL TRIAL: NCT03039075
Title: Comparison of Metformin Hydrochloride Sustained-release Tablet (DuLeNing) and Glucophage in Patients With Type 2 Diabetes
Brief Title: Metformin SR Tablet (DuLeNing) and Glucophage in Patients With Type 2 Diabetes
Acronym: CQM-2016
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qifu Li, Primary Investigator, Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQ-Metformin-2016
Record Dates: First submitted 2016-11-10; First posted 2017-02-01 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin SR Tablet (Active Comparator): Metformin hydrochloride sustained-release tablets made in Conquer pharmaceutical co., LTD
  Interventions: Drug: Metformin SR Tablet
- Glucophage (Active Comparator): The original drug of metformin
  Interventions: Drug: Metformin SR Tablet

INTERVENTIONS:
Drug: Metformin SR Tablet — Metformin SR Tablet made in Conquer pharmaceutical co., LTD
  Other Names: DuLeNing

SUMMARY:
Metformin hydrochloride sustained-release tablets made in Conquer pharmaceutical co., LTD is approved by China Food And Drug Administration (cFDA). Whether its efficacy and safety are equal to Glucophage is unclear.

DETAILED DESCRIPTION:
To perform a RCT for the comparison between Metformin hydrochloride sustained-release tablets made in Conquer pharmaceutical co., LTD and Glucophage .

ELIGIBILITY:
Inclusion Criteria:

1. Well informed of the procedures of this trial and informed consent is obtained
2. Voluntarily accept standardized treatment 3.18-75 years old, gender is not limited

4.Newly diagnosed as type 2 diabetes and have not yet received any hypoglycemic therapy 5.Unable to control the blood glucose by diet and exercise: 7.5% ≤HbA1c ≤11.0%, in screening and before randomization 6.BMI: 19~35 kg/m2 7.Well compliance 8.Capable of self blood Glucose monitoring

Exclusion Criteria:

1. Pregnant or lactating
2. Type 1 diabetes
3. Poor blood glucose control（HbA1c>11%）
4. A history of malignant tumor
5. Abnormal liver or renal function (defined as alanine aminotransferase(ALT)>2.5 times higher than normal range,or eGFR<45 mL/min per 1•73 m²)
6. Poor blood pressure control [systolic blood pressure(SBP)>180mmHg,or diastolic blood pressure(DBP)>110mmHg]
7. With severe heart disease,cardiac function worse than grade II,anemia(Hb<9.0g/d1)
8. Continuous use of antidiabetic drugs more than one week in recent 3 months
9. History of acute metabolic complications in recent 6 months
10. Blood routine test indicates that the white blood cell count(WBC) <3*109/l
11. Body Mass Index(BMI)<18.5 or ≥35kg/m2
12. Drug or alcohol abuse
13. Accompanying mental disorder who can't collaborate
14. Abnormal digestion and absorption function
15. Other endocrine diseases
16. Other chronic diseases needed long-term glucocorticoid treatment
17. With severe infection, immune dysfunction
18. A history of metformin allergies or allergic constitution

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Changes of HbA1c | 12 weeks
  Efficacy

SECONDARY OUTCOMES:
Incidence of nausea, diarrhea | 12 weeks
  Safety
Changes of weight | 12 weeks
Changes of intestinal flora proportion | 12 weeks
Changes of LDL, HDL, TG, TC | 12 weeks
  blood lipid

CONTACTS AND LOCATIONS:
Overall Officials: Qifu Li, phD, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buse JB, DeFronzo RA, Rosenstock J, Kim T, Burns C, Skare S, Baron A, Fineman M. The Primary Glucose-Lowering Effect of Metformin Resides in the Gut, Not the Circulation: Results From Short-term Pharmacokinetic and 12-Week Dose-Ranging Studies. Diabetes Care. 2016 Feb;39(2):198-205. doi: 10.2337/dc15-0488. Epub 2015 Aug 18. PMID 26285584
- [Background] Xu T, Brandmaier S, Messias AC, Herder C, Draisma HH, Demirkan A, Yu Z, Ried JS, Haller T, Heier M, Campillos M, Fobo G, Stark R, Holzapfel C, Adam J, Chi S, Rotter M, Panni T, Quante AS, He Y, Prehn C, Roemisch-Margl W, Kastenmuller G, Willemsen G, Pool R, Kasa K, van Dijk KW, Hankemeier T, Meisinger C, Thorand B, Ruepp A, Hrabe de Angelis M, Li Y, Wichmann HE, Stratmann B, Strauch K, Metspalu A, Gieger C, Suhre K, Adamski J, Illig T, Rathmann W, Roden M, Peters A, van Duijn CM, Boomsma DI, Meitinger T, Wang-Sattler R. Effects of metformin on metabolite profiles and LDL cholesterol in patients with type 2 diabetes. Diabetes Care. 2015 Oct;38(10):1858-67. doi: 10.2337/dc15-0658. Epub 2015 Aug 5. PMID 26251408